CLINICAL TRIAL: NCT03338725
Title: Effect and Associated Factors of the Clinical Pharmacy Model in the Incidence of Medical Errors in the Hospital Pablo Tobon Uribe- Colombia
Brief Title: Effect and Associated Factors of the Clinical Pharmacy Model in the Incidence of Medical Errors
Acronym: EACPharModel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Hospital Pablo Tobón Uribe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0016052017JG
Record Dates: First submitted 2017-10-09; First posted 2017-11-09 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2018-10

CONDITIONS: Pharmaceutical Services; Medication Errors; Drug-Related Side Effects and Adverse Reactions; Outcome Assessment (Health Care)
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trials and The Stepped Wedge (Cluster Analysis Mesh Terms)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without intervention (Active Comparator): Patients without follow-up by clinical pharmacy model
  Interventions: Other: Clinical pharmacy model
- Patients with intervention (Experimental): Patients who are being monitored by a clinical pharmacy model
  Interventions: Other: Clinical pharmacy model

INTERVENTIONS:
Other: Clinical pharmacy model — Patients who are being monitored by a clinical pharmacy model

SUMMARY:
Medication errors are considered by WHO to be a subject that requires attention at all levels of care, in order to reduce the serious and preventable damage related to medication.

These strategies are aimed at the patient's safety policy. In Colombia, at the regulatory level there is no standardized clinical pharmacy model where the role of the clinical pharmacist is described extensively and in detail, and in addition, data are unknown of the scope or direct effect of the incorporation of this model in the assistance in the results of health care.

The Hospital Pablo Tobón Uribe, it is a highly complex institution in Medellin (Colombia), certified by Join Comission International (JCI), which requires the continuous interaction of the pharmacist in patient care, in order to avoid medication errors and contribute to patient safety indicators. In this sense, the hospital structured and implemented a clinical pharmacy model that establishes the activities of the pharmacist incorporated into the care team in the patient attention. Today this model is applied in the institution, however, it is necessary to know the effect of its application in the solution of drug-related problems (DRPs) or a negative outcome related to medicine. The objective of this study is to know the effect on patient safety of a clinical pharmacy model in a hospital of high complexity and framed in the WHO initiative to reduce these errors of medication.

DETAILED DESCRIPTION:
A randomized controlled clinical trial of stepped wedge will be performed. Patients will be admitted according to the inclusion criteria. Randomization will be done at the cluster level (group) and the result measured in the participants within the cluster.

ELIGIBILITY:
Inclusion Criteria:

* To be hospitalized in the Hospital Pablo Tobón Uribe a minimum of 24 hours.
* Patient with at least 5 drugs in their pharmacological therapy

Exclusion Criteria:

* Patients with only surgical procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
The probability of developing medication errors over a certain period of time and recommendations to avoid such errors. | 2 months
  Identify and analyze the types of medication errors

SECONDARY OUTCOMES:
Problems related with the pharmacotherapy | 2 months
  Identify, quantify and classify problems related with the pharmacotherapy:
  If any prescription in a patient have at least on of: Incorrect dosage, Incorrect frequency, Incorrect route of administration, Incorrect duration of therapy, drug not indicated, Contraindicated drug, Lack of treatment, Drug-drug interaction, Drug-food Interaction, Therapeutic duplicity. it is considered as problem related with the pharmacotherapy
  According whit the oficial FDA label of each drug.
Factors that contribute to the occurrence of process and outcomes problems | 2 months
  The factors that influence the occurrence of errors will be estimated through logistic regression
To classify according to the clinical severity the results problems detected | 2 months
  To classify according to the clinical severity the results problems detected:
  A-Circumstances or incidents that are capable of causing error B-The error occurred but did not reach the patient C-The error reached the patient, but did not cause harm D-The error reached the patient and did not cause damage, but needed follow-up to check it E-The error contributed or caused temporary damage to the patient and required intervention F-The error contributed or caused temporary damage and specified or prolonged hospitalization G-The error contributed or caused permanent damage to the patient H-The error affected the life of the patient I-The error contributed or caused the death of the patient
Estimate adjusted survival distribution curves determined by Cox proportional hazards method, in order to estimate the probability that a subject re-mains free of an error medication and its resolution over the time | 14 months
  Estimate adjusted survival distribution curves determined by Cox proportional hazards method, in order to estimate the probability that a subject re-mains free of an error medication and its resolution over the time

CONTACTS AND LOCATIONS:
Overall Officials: Johann Granados, Msc, Principal Investigator — Hospital Pablo Tobon Uribe
Locations (1):
- Hospital Pablo Tobon Uribe, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Granados J, Amariles P, Botero-Aguirre JP, Ortiz-Cano NA, Valencia-Quintero AF, Salazar-Ospina A. Effect and associated factors of a clinical pharmacy model in the incidence of medication errors in the hospital Pablo Tobon Uribe eacpharmodel study: stepped wedge randomized controlled Trial (NCT03338725). Int J Clin Pharm. 2022 Apr;44(2):439-447. doi: 10.1007/s11096-021-01361-9. Epub 2022 Jan 3. PMID 34977994
- [Derived] Granados J, Salazar-Ospina A, Botero-Aguirre JP, Valencia-Quintero AF, Ortiz N, Amariles P. Effect and associated factors of a clinical pharmacy model in the incidence of medication errors (EACPharModel) in the Hospital Pablo Tobon Uribe: study protocol for a stepped wedge randomized controlled trial (NCT03338725). Trials. 2020 Jan 6;21(1):26. doi: 10.1186/s13063-019-3945-8. PMID 31907009